CLINICAL TRIAL: NCT01075126
Title: Depakote Vs. Lithium in African Americans With Bipolar Disorder
Brief Title: Safety Study of Depakote Versus Lithium in African Americans With Bipolar Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: key investigator relocated.
Sponsor: Lawson, William B., M.D., PhD, DFAPA (Individual)
Collaborators: Abbott (Industry)
Responsible Party: Lawson, William B., M.D., PhD, DFAPA., Howard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Abbottdepakote1
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Bipolar Disorder
Keywords: bipolar affective disorder; African American; antimanic; lithium; depakote
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid; Lithium

INTERVENTIONS:
Drug: Depakote
Drug: Lithium

SUMMARY:
It is hypothesized that Depakote will be better tolerated then lithium in treating African Americans with bipolar disorder.

DETAILED DESCRIPTION:
This is a 14 week randomized open study of 50 inpatients or outpatients with bipolar I r II. African American subjects will receive lithium or depakote ER. Measures will be made of psychopathology, reported side effects, and study completers. Measures will also be made of RBC/plasma lithium to determine if this level is better predictive of lithium tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Females must be using a contraceptive
* Understand and sing informed consent
* Meet criteria for DSM IV bipolar I or II
* Must have been receiving treatment with depakote or lithium for at least 4 weeks
* Must not have used illicit substances 48 hours before the study

Exclusion Criteria:

* Not takin g lithium o valproate at time of screening
* Alcohol intoxicated or using drugs of abuse other then cannibis
* Presence of psychotic features
* Participation in clinical trail within 1 month of study
* Female subjects pregnant or nursing
* Serious unstable medical or psychiatric illness
* Uncorrected hypothyroidism or hyperthyroidism
* Seizures without a clear and resolved etiology
* Hypersensitivity or intolerance to lithium or valproic acid
* Treatment with injectable depot neuroleptic less then one dosing interval
* Treatment with reversible MAOI, guanethidine, or guanadrel within i week of study
* Treatment with fluoxetine within 8 weekS of study
* treatment with clozapine or ECT 3 months prior to study
* current diagnosis of schizophrenia or other psychotic disorder
* judged to be at serious suicidal risk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-12; Primary Completion 2006-12 (Estimated); Study Completion 2006-12 (Estimated)

PRIMARY OUTCOMES:
psychopathology: YMRS, MADRS
Tolerability: Uku side effect rating, drop out rate, failure to switch rate

SECONDARY OUTCOMES:
HAMD, CGI-BP, HAM A,CORE, MADRS

CONTACTS AND LOCATIONS:
Overall Officials: William B. Lawson, MD, PhD, Principal Investigator — Professor and Chair, Howard University College of Medicine
Locations (1):
- Howard University Hospital, Washington D.C., District of Columbia, United States